CLINICAL TRIAL: NCT00746863
Title: Injection of 0.125% Marcaine During Mid-Urethral Sling Placement for Pain Relief: A Randomized Control Trial
Brief Title: Randomized Control Trial to Assess Postoperative Pain After Sling Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Gena Dunivan, Clinical Fellow, UNC Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-1890
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Stress Urinary Incontinence
Keywords: mid-urethral sling; pubovaginal sling; postoperative pain; visual analog scale; suprapubic approach; SPARC sling
MeSH Terms: conditions — Urinary Incontinence, Stress; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients randomized to this arm will receive 60 cc of 0.125% Marcaine injected into the retropubic space along the tract that the suprapubic mid-urethral trocar will follow (one on each side) for a total of 120 cc of 0.125% Marcaine, prior to the placement of the mid-urethral sling via the suprapubic approach.
  Interventions: Drug: 0.125% Marcaine
- 2 (No Intervention): Patients assigned to this arm will have the mid-urethral sling placed via the suprapubic approach in the standard fashion with no injection of Marcaine into the retropubic space.

INTERVENTIONS:
Drug: 0.125% Marcaine — Patients randomized to the intervention arm will receive 60 cc of 0.125% Marcaine injected into the retropubic space along the tract that the suprapubic mid-urethral trocar will follow (one on each side) for a total of 120 cc of 0.125% Marcaine, prior to the placement of the mid-urethral sling via the suprapubic approach.
  Other Names: 0.125% Bupivacaine
  Arms: 1

SUMMARY:
There are many ways to perform a suprapubic approach pubovaginal sling. Some surgeons inject local pain medical into the retropubic space before placing the sling, others do not. This study is to determine if injection of local pain medication into the retropubic space before placing a mid-urethral sling for urinary stress incontinence results in lower postoperative pain scores, lower use of postoperative narcotic medication and lower rates of urinary retention.

DETAILED DESCRIPTION:
To evaluate if an injection in the retropubic space with a local acting anesthetic, Marcaine, (bupivacaine) at the time of mid-urethral sling placement will improve patients' reported post operative pain and decrease the use of narcotic pain medication. This study will include all female patients age 18 and older who will undergo a mid-urethral sling with or without anterior repair for the treatment of urinary stress incontinence by a member of the Division of Urogynecology and Reconstructive Pelvic Surgery who consent to be in the study.

Once patients have consented to participate in the study they will be randomized into two groups. One group will have the mid-urethral sling placed in the usual fashion with no injection of local anesthetic. The other group will have the mid-urethral sling placed after the retropubic space has been infiltrated with local anesthetic as previously described in the literature. Pain will be assessed with the use of a Visual Analog Scale during the hospitalization and the use of narcotic pain medication will be assessed during recovery and overnight in the hospital. Patients will be asked to record how often and what type of pain medication they use. Patients will also be asked to keep a log of their urination if they are discharged home with self catheterization. They will be asked to mail in their pain medication log and voiding diary (if needed) at a two-week post-operative. Outcomes will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Any female patient, age 18 or older, who elects to have a mid-urethral sling with or without an anterior or posterior repair at the University of North Carolina Hospitals by a member of the Division of Urogynecology.

Exclusion Criteria:

* Any patient with a chronic pain syndrome, a contraindication to nonsteroidal anti-inflammatory drugs (NSAIDs) such as liver disease, abnormal coagulation, esophageal disorders or peptic ulcers or where pain evaluation is unreliable because of neurological disease and those on treatment with steroids/NSAIDs/opioids prior to surgery.
* Also excluded will be any patient who is having any other reconstructive pelvic surgery concomitantly or would require the placement of a suprapubic catheter.
* Patients electing to have their surgery with regional anesthesia, such as an epidural or spinal will be excluded.
* All minors, decisional impaired people, nursing mothers and non-English speaking people will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gena C Dunivan, MD, Principal Investigator — University of North Carolina, Chapel Hill; Ellen C Wells, MD, Study Director — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Al-Hayek S, Abrams P. Women's lower urinary tract function and dysfunction: definitions and epidemiology. Minerva Ginecol. 2004 Aug;56(4):311-25. PMID 15377981
- [Background] Hunskaar S, Vinsnes A. The quality of life in women with urinary incontinence as measured by the sickness impact profile. J Am Geriatr Soc. 1991 Apr;39(4):378-82. doi: 10.1111/j.1532-5415.1991.tb02903.x. PMID 2010587
- [Background] van der Vaart CH, de Leeuw JR, Roovers JP, Heintz AP. The effect of urinary incontinence and overactive bladder symptoms on quality of life in young women. BJU Int. 2002 Oct;90(6):544-9. doi: 10.1046/j.1464-410x.2002.02963.x. PMID 12230614
- [Background] Leach GE, Dmochowski RR, Appell RA, Blaivas JG, Hadley HR, Luber KM, Mostwin JL, O'Donnell PD, Roehrborn CG. Female Stress Urinary Incontinence Clinical Guidelines Panel summary report on surgical management of female stress urinary incontinence. The American Urological Association. J Urol. 1997 Sep;158(3 Pt 1):875-80. doi: 10.1097/00005392-199709000-00054. PMID 9258103
- [Background] Nilsson CG, Kuuva N, Falconer C, Rezapour M, Ulmsten U. Long-term results of the tension-free vaginal tape (TVT) procedure for surgical treatment of female stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12 Suppl 2:S5-8. doi: 10.1007/s001920170003. PMID 11450979
- [Background] Richter HE, Norman AM, Burgio KL, Goode PS, Wright KC, Benton J, Varner RE. Tension-free vaginal tape: a prospective subjective and objective outcome analysis. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Mar-Apr;16(2):109-13. doi: 10.1007/s00192-004-1238-5. Epub 2004 Oct 23. PMID 15789144
- [Background] Ulmsten U, Henriksson L, Johnson P, Varhos G. An ambulatory surgical procedure under local anesthesia for treatment of female urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):81-5; discussion 85-6. doi: 10.1007/BF01902378. PMID 8798092
- [Background] Schatz H, Henriksson L. Pain during the TVT procedure performed under local anesthesia. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Nov;14(5):347-9; discussion 349. doi: 10.1007/s00192-003-1043-6. Epub 2003 Sep 6. PMID 14618314
- [Background] Dogan E, Celiloglu M, Sarihan E, Demir A. Anesthetic effect of intrauterine lidocaine plus naproxen sodium in endometrial biopsy. Obstet Gynecol. 2004 Feb;103(2):347-51. doi: 10.1097/01.AOG.0000109519.74229.30. PMID 14754707
- [Derived] Dunivan GC, Parnell BA, Connolly A, Jannelli ML, Horton BJ, Geller EJ. Bupivacaine injection during midurethral sling and postoperative pain: a randomized controlled trial. Int Urogynecol J. 2011 Apr;22(4):433-8. doi: 10.1007/s00192-011-1362-y. Epub 2011 Feb 12. PMID 21318442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2008 to September of 2009, all female patients planning to undergo a sling with or without an anterior or posterior repair at the University of North Carolina (UNC) Hospital were approached for participation.
Groups:
- Intervention Group - Received Marcaine: Patients randomized to this arm will receive 60 cc of 0.125% Marcaine injected into the retropubic space along the tract that the suprapubic mid-urethral trocar will follow (one on each side) for a total of 120 cc of 0.125% Marcaine, prior to the placement of the mid-urethral sling via the suprapubic approach.
- Control Group - No Marcaine: Patients assigned to this arm will have the mid-urethral sling placed via the suprapubic approach in the standard fashion with no injection of Marcaine into the retropubic space.
Period: Overall Study
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.5) | 52.6 (10.7) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Only female patients
  Participants
    Female | 21 | 21 | 42
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Difference in Postoperative Pain Using a Visual Analog Scale at 2 Hours.
Description: At approximately two hours postoperatively patients completed a visual analog scale (VAS), which was a 10-cm numeric scale on which 0 represented "no pain" and 10 represented the" worst pain ever".
Time Frame: 2 hours postoperative from mid-urethral sling placement
Population: Analysis was intention to treat. One patient in the intervention did not have a 2 hour VAS collected.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Number analyzed (Participants) | 20 | 21
cm | 1.9 (2.38) | 2.6 (1.78)
Statistical Analysis 1: Comparison: Intervention Group - Received Marcaine vs Control Group - No Marcaine; A 2.0 cm difference on a 10.0 cm VAS scale was clinically significant. Assuming a power of 80% to detect a 2.0 difference on scores between groups, standard deviation of 2.2, an α of 0.05, then, 21 patients would be needed in each group for a total of 42 subjects. A t-test was used in comparing the intervention and control groups, if continuous variables were approximately normal. If data were not approximately normal, a Mann-Whitney Wilcoxon test was used in comparing the two groups; Test type: Superiority or Other; p = 0.0251, Wilcoxon (Mann-Whitney) — A Bonferroni correction was used when evaluating the VAS results to adjust for multiple comparisons

2. Secondary Outcome: In-hospital Medication Amounts
Description: Secondary outcome included differences in amount of pain medication used in the hospital. This was assessed by comparing the number of pills of oral narcotics the patient took while hospitalized.
Time Frame: From surgery until discharge, average
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Number analyzed (Participants) | 21 | 21
number of pills | 4 (3.83) | 6 (4.32)
Statistical Analysis 1: Comparison: Intervention Group - Received Marcaine vs Control Group - No Marcaine; A t-test was used in comparing the intervention and control groups, if continuous variables were approximately normal. If data were not approximately normal, a Mann-Whitney Wilcoxon test was used in comparing the two groups; Test type: Superiority or Other; p = 0.0923, Wilcoxon (Mann-Whitney) — Adjusted for multiple comparisions

3. Secondary Outcome: Difference in Successful Voiding Trial Prior to Discharge Following Placement of Mid-urethral Sling Via the Suprapubic Approach.
Description: Prior to discharge, patients underwent voiding trials. At our institution, in order to pass the voiding trial, they must void at least 200 cc spontaneously and have less than 100 cc as a post void residual two times in a row.
Time Frame: From after surgery to discharge from hospital.
Measure: Number; unit: participants w/sucessful voiding trial
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Number analyzed (Participants) | 21 | 21
participants w/sucessful voiding trial | 4 | 7
Statistical Analysis 1: Comparison: Intervention Group - Received Marcaine vs Control Group - No Marcaine; Chi square was performed to compared the two groups and the patient's ability to pass their voiding trial prior to discharge; Test type: Superiority or Other; p = 0.4756, Chi-squared

4. Primary Outcome: Difference in Postoperative Pain Using a Visual Analog Scale at 6 Hours.
Description: At approximately six hours postoperatively patients completed a visual analog scale (VAS), which was a 10-cm numeric scale on which 0 represented "no pain" and 10 represented the" worst pain ever".
Time Frame: 6 hours postoperative from mid-urethral sling placement
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Number analyzed (Participants) | 21 | 21
cm | 2.1 (2.46) | 2.3 (2.0)
Statistical Analysis 1: Comparison: Intervention Group - Received Marcaine vs Control Group - No Marcaine; A t-test was used in comparing the intervention and control groups, if continuous variables were approximately normal. If data were not approximately normal, a Mann-Whitney Wilcoxon test was used in comparing the two groups. Normality of continuous variables was assessed using the Shapiro-Wilk test. For categorical data, Fisher's exact test was used to evaluate the data. A Bonferroni correction was used when evaluating the VAS results to adjust for multiple comparisons; Test type: Superiority or Other; p = 0.258, Wilcoxon (Mann-Whitney) — A Bonferroni correction was used when evaluating the VAS results to adjust for multiple comparisons

5. Primary Outcome: Difference in Postoperative Pain Using a Visual Analog Scale at 24 Hours.
Description: At approximately twenty-four hours postoperatively patients completed a visual analog scale (VAS), which was a 10-cm numeric scale on which 0 represented "no pain" and 10 represented the" worst pain ever".
Time Frame: 24 hours postoperative from mid-urethral sling placement
Population: Analysis was intention to treat. One patient in the control group was discharged before her 24 hour VAS was collected.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Number analyzed (Participants) | 21 | 20
cm | 2.0 (2.37) | 2.3 (2.22)
Statistical Analysis 1: Comparison: Intervention Group - Received Marcaine vs Control Group - No Marcaine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.435, Wilcoxon (Mann-Whitney) — A Bonferroni correction was used when evaluating the VAS results to adjust for multiple comparisons

ADVERSE EVENTS:
Time Frame: From time of surgery to 6 weeks after surgery
Description: A total of 4 adverse events were documented, 3 in the intervention group and one in the control group. These included right hip pain, a right labial hematoma, a patient with prolonged urinary retention requiring sling release and one blood transfusion. However, these were felt to be related to the surgery itself.
Arm/Group | Intervention Group - Received Marcaine | Control Group - No Marcaine
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 3/21 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group - Received Marcaine (N=21) | Control Group - No Marcaine (N=21)
Blood transfusion (Surgical and medical procedures) | 1 (1) | 0 (0) — One patient in the Intervention group - Marcaine, required a blood transfusion postoperatively secondary to low starting hematocrit preoperatively.
Labial hematoma (Surgical and medical procedures) | 1 (1) | 0 (0) — One patient in the Intervention group - Marcaine, had a labial hematoma noted postoperatively, this self-limited and resolved spontaneously
Hip pain (Surgical and medical procedures) | 1 (1) | 0 (0) — One patient in the Intervention group - Marcaine, complained of right hip pain on postoperative day 1. This resolved with conservative measures.
Prolonged voiding dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1) — One patient in the Control group - No marcaine, had prolonged incomplete emptying and had a release of her sling 6 weeks after her initial surgery.

LIMITATIONS AND CAVEATS:
Our exclusion criteria were strict, and as such, results presented here may have limited generalizability. Other limitations include that we can only address operations performed under general anesthesia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No